CLINICAL TRIAL: NCT03935750
Title: Anterior Cruciate Ligament Reconstruction Using Bone Patellar Bone or Quad Tendon Autograft With or Without Lateral Extra-Articular Tenodesis in Individuals Who Are at High Risk of Graft Failure (STABILITY 2)
Brief Title: STABILITY 2: Anterior Cruciate Ligament Reconstruction +/- Lateral Tenodesis With Patellar vs Quad Tendon
Acronym: STABILITY 2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Western Ontario, Canada (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, James J. Irrgang, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20110331; U01AR076144 (NIH)
Record Dates: First submitted 2019-03-25; First posted 2019-05-02 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament Injury; Anterior Cruciate Ligament Reconstruction; Joint Instability
Keywords: Lateral extra-articular tenodesis; Autografting; Allografting; Bone-Patellar Tendon-Bone Grafting
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Joint Instability | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Intervention Model Description: This trial will randomly assign 1236 ACL deficient patients at high risk of re-injury to anatomic anterior cruciate ligament reconstruction (ACLR) using bone patellar tendon bone (BPTB) or quadriceps tendon (QT) autograft with or without a lateral extra-articular tenodesis (LET) in a 1:1:1:1 ratio.
Who Masked: Outcomes Assessor
Masking Description: All outcome assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BPTB + LET (Experimental): Patients will undergo anterior cruciate ligament reconstruction (ACLR) using a bone patellar bone tendon (BPTB) autograft with lateral extra-articular tenodesis (LET).
  Interventions: Procedure: Anterior cruciate ligament reconstruction (ACLR); Procedure: Lateral extra-articular tenodesis (LET)
- BPTB alone (Active Comparator): Patients will undergo ACLR using a BPTB autograft without LET.
  Interventions: Procedure: Anterior cruciate ligament reconstruction (ACLR)
- QT + LET (Experimental): Patients will undergo ACLR using a quadriceps tendon (QT) autograft with LET.
  Interventions: Procedure: Anterior cruciate ligament reconstruction (ACLR); Procedure: Lateral extra-articular tenodesis (LET)
- QT alone (Active Comparator): Patients will undergo ACLR using a QT autograft without LET.
  Interventions: Procedure: Anterior cruciate ligament reconstruction (ACLR)

INTERVENTIONS:
Procedure: Anterior cruciate ligament reconstruction (ACLR) — All participants will undergo an anatomic ACLR with either a BPTB or QT autograft, as randomized.
Procedure: Lateral extra-articular tenodesis (LET) — Participants randomized to the BPTB or QT arms will be randomized a second time to a LET procedure or no additional surgery.
  Arms: BPTB + LET; QT + LET

SUMMARY:
Anterior cruciate ligament (ACL) rupture is one of the most common musculoskeletal injuries in young individuals, particularly those that are active in sports. Up to 30% of individuals under the age of 20 years suffer a re-injury to the reconstructed ACL. Revision ACLR has been associated with degeneration of the articular cartilage and increased rates of meniscal tears, increasing the risk of post-traumatic osteoarthritis (PTOA), additional surgical procedures, reduced physical function and quality of life. As such, strategies to reduce ACLR failure, particularly in young active individuals, are critical to improving short and long-term outcomes after ACL rupture.

There is ongoing debate about the optimal graft choice and reconstructive technique. Three autograft options are commonly used, including the bone-patellar-tendon-bone (BPTB), quadriceps tendon (QT) and hamstring tendon (HT). Additionally, a lateral extra-articular tenodesis (LET) may provide greater stability to the ACLR; however, its effect on failure rate is unclear and surgery-induced lateral compartment OA is a concern.

To definitively inform the choice of autograft and the need for a LET, this multicenter, international randomized clinical trial will randomly assign 1236 young, active patients at high risk of re-injury to undergo ACLR using BPTB or QT autograft with our without LET.

DETAILED DESCRIPTION:
Anterior cruciate ligament reconstruction (ACLR) is complicated by high failure rates in young, active individuals, which is associated with worse outcomes and higher rates of osteoarthritis (OA). ACLR failure reduces quality of life (QOL) and has substantial socioeconomic costs. Therefore, strategies to reduce ACLR failure are imperative. Lateral extra-articular tenodesis (LET) may provide greater stability; however, its effect on the rate of graft failure remains unclear, and surgically-induced lateral compartment OA is a concern given the potential for over-constraint of the joint.

Many surgeons believe that autograft choice for ACLR, with or without LET, does not affect graft failure. Specifically, bone patella tendon bone (BPTB) autograft has been perceived to be just as good as a hamstring tendon (HT) graft. However, recent meta-analyses suggest that BPTB grafts provide better stability, albeit with greater donor site morbidity. Increasingly, quadriceps tendon (QT) autograft is being used for ACLR with claims of comparable stability to the BPTB graft without the donor site morbidity. However, the effects of a QT on graft failure are unknown. Despite its importance, there has not been an adequately powered study to evaluate if BPTB or QT is superior to the other in terms of graft failure rates, return to sports, donor site morbidity, lateral compartment OA and healthcare costs.

Objectives:

Determine if graft type (QT, BPTB, HT) with or without a LET affects:

* Rate of ACL clinical failure 2 years after ACLR;
* Patient-reported outcomes, muscle function, performance-based measures of function (hop tests, drop vertical jump) and return to sports;
* Intervention-related donor site morbidity, complications and adverse outcomes;
* Cost-effectiveness of ACLR and LET. Approach: This is a multicenter, international, randomized clinical trial that will randomly assign 1236 ACL deficient patients at high risk of re-injury, to an anatomic anterior cruciate ligament reconstruction (ACLR) using a BPTB or QT autograft with or without a LET in a 1:1:1:1 ratio. Data from this study will be combined with data from a recently completed randomized clinical trial comparing ACLR with a hamstring tendon (HT) graft with or without LET.

Randomization will be stratified by surgeon, sex, and meniscal status (normal/repaired v meniscectomy) in permuted block sizes to ensure that any differences in outcome attributable to these factors are equally dispersed between treatment groups. Each site will either use traditional or expertise-based randomization. All randomization will use the web-based application available through the data management center.

Methods to Reduce Biases:

Selection Bias between STABILITY 2 Intervention Groups: We will partially determine eligibility prior to surgery. Once in surgery, all patients will undergo an examination under anesthesia and diagnostic arthroscopy to confirm final eligibility. The surgeon will document evidence of the participant's ineligibility in the surgical report that is discovered during surgery (e.g. partial ACL rupture where an ACLR is not performed, multiple ligament reconstruction, chondral lesion requiring more than debridement). The operative notes for all participants that were consented will be included in the study database. The study quality control monitors will review the evidence provided by the operating surgeon (arthroscopic pictures/video of ACL integrity and chondral status) and recommend that either the participant remain in the study or be withdrawn since they were never eligible.

At the traditional randomization sites, full randomization occurs during surgery following arthroscopic evaluation of eligibility, which already serves to reduce the risk of selection bias. The action of requiring evidence of ineligibility at time of surgery therefore, reduces the risk of sampling bias (applicability) in traditional randomization sites. At the expertise-based randomization sites, where randomization to graft type occurs prior to surgery, this action will prevent unsubstantiated post-randomization withdrawals prior to randomization to LET or no LET, which reduces sampling bias (applicability) and selection bias by avoiding unequal exclusions between the LET/no LET assignment since randomization to LET/no LET occurs after the arthroscopic examination. In summary, having to provide evidence of eligibility at surgery will serve as a deterrent for surgeons declaring eligible consenting patients ineligible during surgery, which serves to reduce the likelihood of sampling and selection bias.

Selection Bias between STABILITY 1 (NCT02018354) and STABILITY 2 Comparisons: STABILITY 1 followed the exact same protocols as are proposed for STABILITY 2 and the two studies will be performed immediately in series; thus, changes in ancillary care and surgeon expertise are unlikely. Consequently, analyses that combine data from STABILITY 1 and STABILITY 2 are unlikely to suffer significant between-study selection biases that are usually a concern for non-randomized comparisons. Further, to evaluate selection bias between the STABILITY 1 and STABILITY 2 samples, the baseline characteristics of the samples will be evaluated to identify any systematic differences between the samples.

Performance Bias, Fidelity & Adherence: Surgeons have agreed upon standardization of aspects of the surgical interventions that could potentially influence outcomes. All other aspects of the surgical interventions are meant to be pragmatic and may vary by surgeon. Aspects allowed to vary are not expected to influence outcome. Further, randomization is stratified by surgeon so that nuance differences by surgeon are balanced between groups. In terms of fidelity, all participating surgeons have the necessary expertise to conduct both surgical procedures (BPTB, QT) if they have elected to participate in traditional randomization. Surgeons who have a preference for or greater skill performing one graft type over the other, will participate in expertise-based randomization and have identified another surgeon with similar expertise/preference performing the opposite graft type. In terms of performing a LET, all surgeons who have not completed at least 10 LETs will participate in a cadaver training lab and be required to complete at least 10 LET procedures prior to randomizing their first patient. The investigators have agreed upon a protocol for ACL rehabilitation following ACLR. All patients will receive a copy of the protocol with a standardized referral from their surgeon for their physical therapist. Deviations from the protocol are not expected to be different from usual practice and as such patient adherence with rehabilitation protocols is expected to vary. Given the large sample size, we expect that adherence to rehabilitation will be balanced between groups and we will adjust the analyses for length of time in rehabilitation. This study will track the number of rehabilitation sessions attended, milestones and timing of rehabilitation-specific activities to collect some adherence and fidelity data.

Detection Bias: An independent surgeon, primary care sports medicine physician, physical therapist or athletic trainer who is unaware of group allocation will conduct all assessments of graft stability (primary outcome). Although incisions are unique for each procedure, patients will wear a tubigrip sleeve over both knees to conceal the incisions and reduce bias in assessments that require side-to-side comparisons, including the primary outcome. Data assessors for other outcomes will also be kept unaware of group allocation using this method.

Intention-to-Treat Principle: Patients will be analyzed within the group to which they were randomized regardless of graft type received or adherence to protocols.

Attrition Bias: From STABILITY 1, we have complete data on 95% of the 618 patients who are at least 2 years postoperative demonstrating that we are capable of successful recruitment and retention in a study of this magnitude. We will use the same measures to maximize completeness of follow-up

Statistical Methods:

Sample Size: We estimate that the absolute risk of graft failure (as defined above) in the ACLR will range from 25-35%. STABILITY 1 supports this estimate. We consider a relative reduction in graft failure rate of at least 40% to merit a change in practice (i.e. of sufficient magnitude to warrant the additional costs of adding a LET). With 255 patients per group and a type I error rate of 1% we would have 80% power to detect a relative risk reduction in rate of failure of 40% or greater in those with LET assuming the graft failure rate in ACLR is 33%. We have used a small type I error rate of 1% to reduce the risk of multiple comparisons error. To reduce the risk of losing precision from withdrawal and lost-to-follow-ups, we will over recruit by 15%, for a total of 309 per group or 1853 participants in total (combined STABILITY 1 and STABILITY 2 data).

While not all sites have the infrastructure to conduct the isokinetic quadriceps and hamstring tests (13 sites) and in vivo kinematics during the DVJ (one site), these outcomes are reported using a continuous metric and therefore do not require as large a sample size as the proportional primary outcome.

Statistical Analyses: The data collected through this study will be pooled with the data from STABILITY 1 for analysis (n=1800). To determine whether graft type (QT, BPTB, HT) with or without a LET offers a greater reduction in rate of failure following ACLR (primary research question), we will use a random-effects logistic regression with failure following ACLR at each visit (yes/no) as the outcome where fixed effects include intervention group, meniscal repair status, sex and time (as a categorical variable) and random effects include patient and surgeon. We will conduct a similar analysis for secondary outcomes like return-to-activity and donor site adverse events, as both are binary outcomes. For each continuous secondary outcome including patient-reported outcomes (PRO) scores, measures of impaired range of motion (ROM) and muscle strength, performance-based measures of physical function, and lateral compartment joint space narrowing, we will conduct a linear mixed-effects model where the fixed effects include ACLR group, meniscal repair status, sex and time (as a categorical variable) and random effects including patient and surgeon. For missing data, we will evaluate whether data are missing completely at random by comparing the available data (especially at baseline) for those with and without missing data at follow-up. We will use multiple imputation techniques to handle missing data.

Sex-based analysis: To compare failure between HT+LET and other graft options (BPTB or QT) for males and females separately, we will conduct a random-effects logistic regression with the same fixed and random effects as in the primary analysis.

Health services analyses: We will assign the average procedure cost for an ACLR surgery at each participating institution with the additional cost of the lateral extra-articular tenodesis for those patients randomized to the LET group. Patients who undergo a revision ACLR will complete a healthcare resource diary to capture additional direct and indirect costs. We will conduct a cost-effectiveness analysis from a healthcare payer and societal perspective using quality-adjusted life years (QALY) as our effectiveness outcome at two years postoperative. We will estimate the incremental net benefit (INB) of ACLR + LET using a random effects multilevel model. To characterize the statistical uncertainty around our estimate of INB, we will use an extension of the standard net benefit regression framework using the hierarchical data to generate location-specific net benefit curves, and cost-effectiveness acceptability curves.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-25,
* An ACL-deficient knee,
* Skeletal maturity (i.e. closed epiphyseal growth plates on standard knee radiographs),
* At least two of the following: participate in a competitive pivoting sport; have a pivot shift of grade 2 or greater; have generalized ligamentous laxity (Beighton score of ≥4) and/or genu recurvatum >10 degrees.

Exclusion Criteria:

* Previous ACLR on either knee,
* Partial ACL injury (defined as one bundle ACL tear requiring reconstruction/augmentation of the torn bundle with no surgery required for the intact bundle),
* Multiple ligament injury (two or more ligaments requiring surgery),
* Symptomatic articular cartilage defect requiring treatment other than debridement,
* >3 degrees of asymmetric varus,
* Inflammatory arthropathy,
* Inability to provide consent,
* Pregnancy at baseline.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1236 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
ACL Clinical Failure | 24 months
  This is a composite endpoint defined as 1) graft rupture or, 2) persistent rotational laxity (asymmetrical positive pivot shift).

SECONDARY OUTCOMES:
ACL-Quality of Life (QOL) Questionnaire | 24 months (at 1.5, 3, 6, 12 and 24 months)
  The ACL Quality of Life (QOL) Questionnaire is a patient-reported disease-specific measure of physical symptoms, occupational concerns, recreational activities, lifestyle, social and emotional aspects of ACL injury. Each item has a 0-100 mm visual analogue scale response option (0 represents extremely difficult and 100 not difficult at all). Score is calculated as the average of each item for a total average score out of 100%, where 100% represents the best possible score.
Knee injury and Osteoarthritis Outcome Score (KOOS) | 24 months (at 1.5, 3, 6, 12 and 24 months)
  The Knee injury and Osteoarthritic Outcome Score (KOOS) is a patient-reported knee-specific that consists of 42 items in 5 domains (pain, other symptoms, function of daily living, function in sports/recreation and knee-related quality of life). Each domain is scored by summing the responses of the items in the domain standardized to a score from 0 to 100 (worst to best).
International Knee Documentation Committee Subjective Knee Form (IKDC-SKF) | 24 months (at 1.5, 3, 6, 12 and 24 months)
  The IKDC-SKF is an 18-item questionnaire that assesses symptoms, function and sports activities. The score is calculated by summing the item responses and normalizing to a scale that ranges from 0 to 100 with 100 representing no symptoms or limitations with function and sports activities.
Marx Activity Rating Scale | 24 months (at 1.5, 3, 6, 12 and 24 months)
  The Marx Activity Rating Scale will be used to measure sports activity level. It is a 4-item scale that measures how often patients are able to perform different activities (e.g. running, cutting, decelerating, and pivoting) on a 5-point scale (0 to 4). Scores range from 0 to 16, and higher scores represent higher level of activity.
Side-to-side difference in knee range of motion | 24 months (at 1.5, 3, 6, 12 and 24 months)
  Bilateral passive knee extension and active-assisted knee flexion will be measured with a standard goniometer. The side-to-side difference in range of motion will be calculated and interpreted based on the IKDC guidelines (normal: side-to-side difference in knee extension < 3 degrees and side-to-side difference in knee flexion < 5 degrees; nearly normal or worse).
Isokinetic Quadriceps Strength | 6, 12 and 24 months
  Bilateral quadriceps strength will be measured using a computerized isokinetic dynamometer (assessing maximal concentric torque at an angular velocity of 90°/s). The ratio of peak torque of the involved to non-involved knee will be calculated.
Isokinetic Hamstring Strength | 6, 12 and 24 months
  Bilateral hamstring strength will be measured using a computerized isokinetic dynamometer (assessing maximal concentric torque at an angular velocity of 90°/s) . The ratio of peak torque of the involved to non-involved knee will be calculated.
Isometric Quadriceps Strength | 6, 12 and 24 months
  Bilateral quadriceps strength will be measured using hand-held dynamometer (assessing isometric maximal contraction at 90° of knee flexion). The ratio of peak torque of the involved to non-involved knee will be calculated.
Isometric Hamstring Strength | 6, 12 and 24 months
  Bilateral hamstring strength will be measured using hand-held dynamometer (assessing isometric maximal contraction at 90° of knee flexion). The ratio of peak torque of the involved to non-involved knee will be calculated.
Limb Symmetry Index - Hop test | 6, 12 and 24 months
  Calculated based on the average of four hop tests (single leg hop, 6m timed hop, triple hop, and triple crossover hop). For the single hop for distance, triple hop and triple crossover hop the limb symmetry index (LSI) will calculated as the ratio of the distance hopped on the ACL reconstructed lower extremity to the distance hopped contralateral lower extremity times 100%. For the 6m timed hop, the LSI will be calculated as the ratio of the time to hop 6m on the contralateral normal extremity to the time to hop 6 m on the ACL reconstructed extremity. For analysis, we will use the average of the LSIs for the four hop tests.
Drop vertical jump (DVJ) testing | 6 and 12 months
  The drop vertical jump test will be quantified using a Microsoft Kinect V2 sensor and ACL Gold software to measure dynamic knee valgus that will be defined as the ratio of the distance between the knees to the distance between the ankles. The average ratio of the distance between the knees to ankles across 3 trials will be calculated and use for analysis.
Donor site morbidity - Sensory Disturbance | 24 months (at 1.5, 3, 6, 12 and 24 months)
  Sensory disturbance will be assessed via light touch to regions around the graft skin incision and anterolateral tibia. It will be rated as absent, mild, moderate or severe. This outcome will be presented as the proportion of individuals in each category.
Donor site morbidity - Anterior Kneeling Pain | 24 months (at 1.5, 3, 6, 12 and 24 months)
  Anterior kneeling pain measured using an 11-point numeric rating scale (0 - no pain; 10 - worst imaginable).
Adverse events | 24 months (at 1.5, 3, 6, 12 and 24 months)
  Defined as any new event not present during the pre-intervention period or an event present pre-intervention that has increased in severity.

CONTACTS AND LOCATIONS:
Overall Officials: James J Irrgang, PT PhD FAPTA, Principal Investigator — University of Pittsburgh; Alan Getgood, MD FRCS, Principal Investigator — Fowler Kennedy Sport Medicine Clinic, Western University, Department of Surgery; Volker Musahl, MD, Principal Investigator — University of Pittsburgh; Dianne M Bryant, PhD, Principal Investigator — Western University, School of Physical Therapy & Department of Surgery
Locations (31):
- United States (14):
  - Stanford University, Redwood City, California
  - University of California, San Francisco, San Francisco, California
  - Orlando Health Jewett Orthopedic Institute, Orlando, Florida
  - Med Center Health, Bowling Green, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of New Mexico, Albuquerque, New Mexico
  - Hospital for Special Surgery, New York, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - The Rector and Visitors of the University of Virginia, Charlottesville, Virginia
- Canada (9):
  - Banff Sport Medicine Clinic, Banff, Alberta
  - University of Calgary Sport Medicine Centre, Calgary, Alberta
  - Fraser Health Authority, New Westminster, British Columbia
  - Pan Am Clinic, Winnipeg, Manitoba
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Fowler Kennedy Sport Medicine Clinic, London, Ontario
  - University of Ottawa, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- Aarhus University Hospital, Aarhus, Denmark
- Germany (2):
  - Cologne-Merheim Medical Center, Klinik für Orthopädie, Unfallchirurgie und Sporttraumatologie, Cologne
  - University Klinik Münster, Münster
- Dublin City University / UPMC Sports Surgery Clinic, Dublin, Dublin 9, Ireland
- Oslo University Hospital, Oslo, Norway
- Stockholm South Hospital, Karolinska Institutet, Stockholm, Sweden
- United Kingdom (2):
  - North Bristol Trust, Bristol
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry

IPD SHARING:
Plan to Share IPD: Yes
A public-use version of the dataset will be constructed by the Data Coordinating Center (DCC) with contents to be determined jointly by the study PIs and the DCC Director. Copies of the public-use version of the dataset will be housed at the DCC on the DA secure server along with suitable documentation of this dataset. The public-use version of the dataset will be exported by CRF in one or more files in simple, widely-accessible formats, e.g., .xls, .csv, and/or SAS datasets. Documentation will be in .pdf files.
Supporting Information: Study Protocol
Time Frame: The public-use version of the database will be made available two years after the study's main paper is published.
Access Criteria: Outside investigators wishing to conduct analyses using the data will submit a request with objectives, methods, and analysis plan to the PI and the Director of the DCC. Once the request is approved, the public-use version of the dataset, with documentation, will be sent by secure email using e-mail, ftp, or other mutually agreeable transmission method.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT03935750/Prot_SAP_000.pdf
  • Informed Consent Form (2025-10-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT03935750/ICF_001.pdf